CLINICAL TRIAL: NCT06869057
Title: Re-Engineered Discharge for Diabetes Care Transitions: Screening and Addressing Social Determinants of Health Needs at Hospital Discharge
Brief Title: Re-Engineered Discharge for Diabetes Care Transitions
Acronym: REDDCAT2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Regents of the University of Michigan (Unknown)
Responsible Party: Principal Investigator, Suzanne Mitchell, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002129; R01NR021826 (NIH)
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus Type 2; Social Determinants of Health (SDOH); Hospital Readmission
Keywords: diabetes; social determinants of health; hospital readmission
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Treatment as usual (TAU)
  Interventions: Other: Treatment as Usual (TAU)
- Intervention (Experimental): REDDCAT2 Intervention
  Interventions: Behavioral: REDDCAT2 Post-Discharge Navigation

INTERVENTIONS:
Behavioral: REDDCAT2 Post-Discharge Navigation — Those in the REDDCAT2 intervention group will be partnered with a patient navigator whose role will be to review the results of the screening survey completed at the beginning of the study. The patient navigator will help coordinate the participant's care before leaving the hospital and for 90 days after. Together, the participant and navigator will form an action plan intended to help address personal, social, or community factors affecting the participant's health. The navigator is expected to contact the participant every 2 weeks, though this can be adjusted based on their preference.
  Arms: Intervention
Other: Treatment as Usual (TAU) — TAU participants will receive standard care from the UMass Memorial Healthcare (UMMH) hospitalist team as appropriate. Participants will receive a printed list of community resources. No study-related patient navigation support will be provided.
  In 2024, Centers for Medicare and Medicaid Services mandated social determinants of health (SDOH) screening for inpatients. UMMH will use a checklist social needs screener. It will be up to the hospitalist teams to act on SDOH screening results. The UMMH hospitalist teams may consult endocrinology and/or inpatient social services to provide support and consultation for all patients regardless of study participation or group assignment. If medically appropriate, the endocrinology service may manage medications and provide referrals for continued treatment post discharge. All services that are normally provided by hospital care teams will remain available.
  Arms: Control

SUMMARY:
The goal of this project is to test a novel bedside SDOH screening intervention coupled with post-discharge navigation for hospitalized patients with a diabetes diagnosis to reduce unmet social needs, compared to usual care.

DETAILED DESCRIPTION:
The investigators are conducting this research to test a computer-based screening tool and a care coordination protocol to help people with type 2 diabetes who report unmet social determinants of health.

Social determinants of health (SDOH) are the conditions in the environments where people are born, live, learn, work, play, worship, and age that affect a wide range of health, functioning, and quality-of-life outcomes and risks. - Office of Disease Prevention and Health Promotion Examples of SDOH include factors such as housing, transportation, education, job opportunities, income, and access to healthy food, clean air and water, and health care services. Participants who join this research will be asked to complete a screening survey about their health. Then, participants will be randomly assigned (like pulling a name out of a hat) to one of two groups:

* Those in Group 1 will be partnered with a patient navigator whose role will be to review the results of the screening survey and help coordinate care before leaving the hospital and for 90 days after.
* Those in Group 2 will receive treatment as usual. A list of community-based resources will be provided.

Participants in both groups will complete surveys at the beginning of the study and again at 30 and 90 days after leaving the hospital. The investigators will make reminder calls to participants in both groups about data collection and will collect information from the medical record for as long as 90 days after leaving the hospital.

ELIGIBILITY:
Inclusion Criteria:

* adult aged 18 years or older
* diagnosed with type 2 diabetes
* hospitalized at Univ of Massachusetts-affiliated hospital
* endorsed at least 1 unmet social need via screening survey

Exclusion Criteria:

* pregnancy
* discharge to short or long-term nursing facility or hospital
* medical contraindication
* cognitive impairment
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Time to hospital service use post-discharge | 90 days
  The primary outcome is a composite measure on all types of hospital service use (emergency department, observation, or hospital readmissions), pre-specified as time-to-hospital reutilization, at 90-days post-hospital discharge. Source of the data are UMMH electronic health records and participant self-report.

SECONDARY OUTCOMES:
Changes in weight/body mass index (BMI) | Baseline, 30, and 90 days
  Change in weight/BMI per electronic health record or Research Assistant assessment
Changes in Pain Management | Baseline, 30, and 90 days
  Change in Pain and Pain interference scores assessed using two measures from the Patient-Reported Outcomes Measurement Information System (PROMIS).
  1. Pain Severity is scored using a T-score ranging from 20 to 80. T-scores that are 1 or more standard deviations above average are indicative of a poorer outcome (more pain).
  2. Pain Interference, which is a T-score ranging from 20 to 80. T-scores that are 1+ standard deviations above average are indicative of a poorer outcome (more problems with pain hindering activities).
  PROMIS scores have an average of 50 and standard deviation (SD) of 10 in a referent population.
Changes in Self-Management Adherence | Baseline, 30, and 90 days
  Change in patient-reported adherence to diabetes regimen from baseline to follow up assessed by administering the Changes in the Summary of Diabetes Self-Care Activities Assessment (SDSCA) & Re-Engineered Discharge for Diabetes Computer Adaptive Test (REDD-CAT) for Medication Adherence.
  SDSCA - Scores are calculated for each of the five regimen areas assessed: Diet, Exercise, Blood-Glucose Testing, Foot Care, and Smoking Status.
  REDD-CAT Medication Adherence scale is measured using T-scores. Scores greater that 1 standard deviation of 10.0 away from the mean of 50.0 represent a greater or lesser degree of adherence, depending on direction. Higher scores are indicative of a positive outcome (more adherence).
Changes in Illness Burden perception | Baseline, 30, and 90 days
  Change in experience of Illness Burden. Illness burden scale generates a T-score, ranging from 20 to 80. The average score is 50 with a standard deviation of 10. T-scores that are 1 or more standard deviations above average are indicative of a poorer outcome (indicate more illness burden).
Changes in Substance Use | Baseline, 30, and 90 days
  Change in Substance Use will be assessed using a validated measure from the Patient-Reported Outcomes Measurement Information System (PROMIS). PROMIS scores have an average of 50 and standard deviation (SD) of 10 in a referent population.
  PROMIS Substance Use - Resulting scores are on a T-score metric ranging from 20 to 80. Scores that are 1 or more standard deviations above average are indicative of poor, self-reported health (greater severity of substance use).
Changes in Alcohol Use | Baseline, 30, and 90 days
  Change in Alcohol Use will be assessed using a validated measure from the Patient-Reported Outcomes Measurement Information System (PROMIS). PROMIS scores have an average of 50 and standard deviation (SD) of 10 in a referent population.
  PROMIS Alcohol Use: Resulting scores are on a T-score metric ranging from 20 to 80. Higher scores are indicative of poor self-reported health (more alcohol consumption, cravings, or difficulty controlling drinking).
Changes in Diabetes Stigma | Baseline, 30, and 90 days
  Type 2 Diabetes Stigma Assessment Scale or DSAS-2 is a 19-item measure with three sub-scales: Treated Differently, Blame and Judgement, Self-Stigma. A total scale score can also be calculated. Items are scored 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate worse outcomes (more perceived diabetes stigma).
Changes in Economic Quality of Life | Baseline, 30, and 90 days
  Changes in 8-item custom short form from the Economic Quality of Life item bank. Items are related to finances and affordability of living expenses and range from 1 (Never) to 5 (Always). Resulting scores are on a T-score metric, ranging from 20 to 80. Higher scores indicate better economic quality of life.
Changes in Depressive Symptoms | Baseline, 30, and 90 days
  Changes in depressive symptom burden are assessed using a measure from the Quality of Life in Neurological Disorders (NeuroQOL) measurement system.
  Neuro-QoL Depression - Resulting scores are on a T-score metric, ranging from 20 to 80. Higher scores indicate poorer self-reported health (a greater presence of depressive symptoms).
Changes in Anxiety Symptoms | Baseline, 30, and 90 days
  Changes in anxiety symptom burden are assessed using a measure from the Quality of Life in Neurological Disorders (NeuroQOL) measurement system.
  Neuro-QoL Anxiety - Resulting scores are on a T-score metric, ranging from 20 to 80. Higher scores indicate poorer self-reported health (a greater presence of anxiety symptoms).
Changes in Emotional Support | Baseline, 30, and 90 days
  Changes in emotional support scores assessed using measures from the Patient-Reported Outcomes Measurement Information System (PROMIS).
  Resulting scores are on a T-score metric, ranging from 20 to 80. Higher scores indicate worse outcome (a greater degree of social isolation).
Changes in Health Seeking Behavior | Baseline, 30, and 90 days
  Changes in Health Seeking Behavior scale, which includes 21 items including subscales related to Primary Care Provider, General, Family/Personal Friends, and Internet. Resulting scores are on a T metric, ranging from 20 to 80. Higher scores indicate a positive outcome (more health-seeking behavior).
Changes in Medication Adherence | Baseline, 30, and 90 days
  Medication Adherence scores assessed by administering the Re-Engineered Discharge for Diabetes Computer Adaptive Test (REDD-CAT) for Medication Adherence scale.
  This is measured using T-scores. Scores greater that 1 standard deviation of 10.0 away from the mean of 50.0 reflect a greater or lesser degree of adherence, depending on direction. Higher scores are indicative of a positive outcome (more adherence).
Changes in Perceived Competence | Baseline, 30, and 90 days
  Change in Perceived Competence in Diabetes Scale (PCDS) score - items are rated on a scale 1-7. Higher total scores indicate better self-reported health (a greater perceived ability to manage diabetes).
Changes in Perceived diabetes self-efficacy | Baseline, 30, and 90 days
  Change in Diabetes Self-Efficacy Scale (DSES) score - items are rated on a scale of 0-10 and summed for a total score. Higher total scores indicate better self-reported health (self-efficacy in managing diabetes).
Changes in Coping Skills | Baseline, 30, and 90 days
  Changes in Brief Resilient Coping Scale scores. Items are rated 1 ("does not describe me at all") to 5 ("describes me very well") and summed for a total score. Higher scores indicate better self-reported health (higher coping resiliency).
Changes in Diabetes Knowledge | Baseline, 30, and 90 days
  Change in Diabetes Knowledge and diabetes self-care will be assessed using the 23-item Revised Diabetes Knowledge Test (DKT2). DTK2 contains multiple choice questions to assess knowledge, and each question contains 4 responses for the respondent to choose from. Proportion of correct answers over total questions determine scoring.
Changes in Housing Insecurity | Baseline, 30, and 90 days
  Change in Housing Insecurity scores, which is a 22-item assessment to evaluate affordability, safety, and home features. Resulting scores use a T-score metric, ranging from 20 to 80. Lower scores indicate poorer outcomes (more significant concerns with housing stability).
Quantity of unmet social needs | Baseline, 30, and 90 days
  Absolute change in total number of SDOH domains identified with an unmet need (i.e., food insecurity, housing insecurity, etc.) as reported on Re-Engineered Discharge for Diabetes Computer Adaptive Test (REDD-CAT) screening tool.
Changes in Glucose Control: HbA1c at point of care | Baseline and 90 days
  Change in HbA1c values recorded from point-of-care tests or in the electronic health record at visits.
changes in Diabetes Distress | Baseline, 30, and 90 days
  The Diabetes Distress Scale is a 17-item self-report instrument. Each item is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem." The scale yields an overall distress score based on the average responses on the 1-6 scale for all 17 items. The scale also yields a score for each of 4 subscales based on the average response on the 1-6 scale on all of the items in that scale.
  An average score of < 2.0 = reflects little or no distress, an average score between 2.0 and 2.9 = reflects moderate distress, and an average score > 3.0 = reflects high distress.
Time to hospital service use post-discharge | 30 days
  Time-to-hospital reutilization (defined as any type of hospital service use, e.g., emergency department, observation, or hospital readmissions), at 30-days post-hospital discharge. Source of the data are UMMH electronic health records and participant self-report.

IPD SHARING:
Plan to Share IPD: No
This is a clinical trial. We plan to share data in aggregate according to our data management sharing plan. Sharing individual-level data is beyond the scope of this study.

DOCUMENTS (1):
  • Informed Consent Form (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT06869057/ICF_000.pdf